CLINICAL TRIAL: NCT07189494
Title: ENSEMBLE: European Newborn Study: Early Markers for a Better LifE
Brief Title: European Newborn Study: Early Markers for a Better LifE
Acronym: ENSEMBLE
Status: Recruiting | Type: Observational
Sponsor: dr. M.J.N.L. Benders (Other)
Collaborators: Fondation Paralysie Cérébrale (Other); Zoundream (Unknown); CP Nederland (Unknown); NeuroSpin (Unknown)
Responsible Party: Sponsor-Investigator, dr. M.J.N.L. Benders, Prof. dr., UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: NL83183.041.22
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; machine learning; diagostic tool
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to create a computer model to help doctors predict any problems occurring during development of babies after being diagnosed with brain injury. This will help provide better care to future babies. Next to this, the experiences of parents or caregivers surrounding the first two years after birth of a baby at risk of developing cerebral palsy will be researched to develop recommendations to support parents.

Parents of participants will:

- Fill in two online questionnaires, one when their child is 3-4 months corrected age. The second when their child is 2 years corrected age.

For the child no additional tests are needed. Only tests that are part of standard clinical practice are performed and are also saved in the study database.

ELIGIBILITY:
Inclusion Criteria:

* All infants with confirmed brain injury on MRI at high risk for CP.

Particularly, infants with the following brain injuries at risk for CP will be considered on MRI at term equivalent age or within 10 days after birth or sentinel event:

* Extensive punctate white matter injury.
* Periventricular hemorrhagic infarction (any location).
* Cerebellar injury (ischemic and/or hemorrhages) involving the vermis or involving more than 1/3 of the cerebellar hemisphere and/or lesions involving the cerebellar vermis (Meijler & Steggerda, 2019).
* Cystic periventricular leukomalacia (grade 3 & 4).
* intraventricular hemorrhages grade III.
* Posthemorrhagic ventricular dilatation exceeding the 97°percentile + 4mm for the ventricular index (Cizmeci et al., 2020).
* Perinatal asphyxia with hypoxic ischemic injury of the central gray matter and/or perirolandic area.
* Perinatal asphyxia with hypoxic ischemic injury in the watershed areas.
* Perinatal ischemic arterial stroke at high risk for CP, thus with involvement of the corticospinal tracts, cortex, white matter and basal ganglia (Wagenaar et al., 2018).
* Presence of other brain injuries with expected adverse motor outcome (i.e. big subdural and parenchymal bleedings with/without midline shift, bilirubin induced brain injury) in preterm infants, term infants with neonatal encephalopathy with/without neonatal seizures.

  * Written informed parental consent (Dutch, English, French, German, Italian, Spanish).

Exclusion Criteria:

* Infants not matching the inclusion criteria.
* Any proven or suspected severe congenital anomaly, genetic or metabolic disorder.
* Presence of an infection of the central nervous system.
* Parents < 18 years old.
* Not being able to read one of the six Informed Consent languages.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include all preterm and term born infants with any brain injury at risk for CP admitted to the neonatal intensive of 8 large European NICUs, high and medium care units, including their parents. Based on a conservative estimate and taking into account incidence of in/exclusion criteria, we expect to include 1000 eligible patients in a total inclusion period of 2.5 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Development of a machine learning based prediction model | Neurodevelopmental outcome at 2 years predicted by clinical data from birth to 3-4 months corrected age
  To develop and evaluate a new prediction model using machine learning to predict the risk, severity, and long-term outcome of cerebral palsy (CP) at the level of the individual patient. This model will also provide automatic scoring for each clinical modality (MRI, EEG, GM, HINE, infant cry), which is to be compared with the clinician assessments.

SECONDARY OUTCOMES:
Gaining insight into parental mental well-being and family= and social functioning. | Parent experience asked in questionnaires at age 3-4 months and 2 years.
  To gain insight in parental mental well-being and family- and social functioning, over the first two years after the birth of their child with brain injury, born preterm or full-term, at high risk of developing CP. Including evaluation of parents' experiences around the disclosure of diagnosis, and the impact of these experiences, child-related factors and social support on parental mental well-being. To understand the needs and preferences of parents on the process of disclosure of diagnosis and on information regarding prediction and prognosis, and to identify what information is meaningful to families.

CONTACTS AND LOCATIONS:
Locations (8):
- Assistance Publique Hôpitaux de Paris, Paris, France
- University Hospital Essen, Essen, Germany
- Italy (4):
  - Ospedale Pediatrico Meyer Firenze, Florence
  - Istituto Giannina Gaslini, Genova
  - Ospedale Maggiore di Milano, Milan
  - Fondazione Stella Maris, Pisa
- UMC Utrecht, Utrecht, Netherlands
- University Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes